CLINICAL TRIAL: NCT00868673
Title: The Role Of Fructose and Uric Acid In the Development of Obesity and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: MD Magdalena Madero R., Instituto Nacional de Cardiología Ignacio Chávez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: FRUCTOSE 09-630
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2009-11

CONDITIONS: Overweight and Obesity; Metabolic Syndrome; Hyperuricemia
Keywords: Role of Fructose in overweight and obesity; Fructose and metabolic syndrome; Low fructose diet study; Effects of fructose in blood pressure and hypertension; Somatometry changes observed in fructose diets; Fructose induced overweight and obesity; Fructose induced metabolic syndrome; Fructose induced hyperuricemia
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Hyperuricemia; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low fructose arm (Active Comparator): Overweighted or obese previously healthy adults (with no other comorbidities, defined as: Diabetes (DM1 or DM2), hypertension, chronic kidney disease (CKD), hepatic damage, dyslipidemia medication, anemia, malignancy or pregnancy), with a Body Mass Index (BMI) of >25 kilograms(weight)/ squared meters (height).
  They will be randomized to a 1500, 1800 or 2000 kilocalories diet calculated by Harris Benedict equation, thermic effect of foods and rest energy (without exercise).
  This group will be assigned to a 2 week period of low fructose diet (less than 10 grams/day ) followed by a 4 week period of less than 20 grams/day fructose diet levels.
  Total Time of intervention 6 weeks for each patient
  Interventions: Dietary Supplement: low fructose
- Normal fructose arm (Active Comparator): Overweighted or obese previously healthy adults (with no other comorbidities; defined as: Diabetes Mellitus (DM1 or DM2), hypertension, chronic kidney disease (CKD), hepatic damage, dyslipidemia medication, anemia, malignancy or pregnancy), with a Body Mass Index (BMI) of >25 kilograms(weight)/ squared meters (height).
  Participants will be randomized to a 1500, 1800 or 2000 kilocalories diet (of 15% proteins, 30% lipids and 55% carbohydrates); calculated by Harris Benedict equation, thermic effect of foods and energy (without exercise).
  This group will receive a controlled fructose diet between 50 and 70 grams/day of fructose intake.
  Total time of intervention:6 weeks for each patient
  Interventions: Dietary Supplement: Normal fructose arm

INTERVENTIONS:
Dietary Supplement: low fructose — patients will receive a low fructose diet to evaluate possible changes in weight loss after a 6 week period of receiving a caloric intake (proteins, fats and carbohydrates) based on their healthy-desired weight. Participants will be randomized to a 1500, 1800 or 2000 kilocalories diet calculated by Harris Benedict equation, thermic effect of foods and energy (without exercise). low fructose arm: a 2 week period of low fructose diet (less than 10 grams/day ) followed by a 4 week period of "healthy" fructose diet levels (less than 20 grams/day).Baseline measurements and weekly monitoring of somatometry parameters (BMI, %body fat, waist and hip Index, blood pressure), lipid profile and uric acid levels will be done.
  Arms: Low fructose arm
Dietary Supplement: Normal fructose arm — patients will receive a normal fructose diet to evaluate possible changes in weight loss after a 6 week period of receiving a caloric intake (proteins, fats and carbohydrates) based on their healthy-desired weight. Participants will be randomized to a 1500, 1800 or 2000 kilocalories diet calculated by Harris Benedict equation, thermic effect of foods and energy (without exercise). Normal fructose arm: participants will receive a 6 week period of normal fructose diet between 50 to 70 grams/day. Baseline measurements and weekly monitoring of somatometry parameters (BMI, %body fat, waist and hip Index, blood pressure), lipid profile and uric acid levels will be done.
  Other Names: NORMAL FRUCTOSE
  Arms: Normal fructose arm

SUMMARY:
The purpose of this study is to determine if a low fructose intake could have an impact on weight loss, uric acid levels and the components of the metabolic syndrome (glucose, cholesterol, triglycerides, insulin resistance, high blood pressure).

DETAILED DESCRIPTION:
Overweight and obesity are now considered a growing public health problem in Mexico and worldwide. This epidemic has been attributed to dietary fructose consumption. Although experimental models have demonstrated a role of fructose in the development of obesity, metabolic syndrome and kidney disease, data in human models is lacking. The purpose of this study is to determine if a low fructose intake could have an impact on the components of the metabolic syndrome. The primary endpoint will be to determine the impact of low fructose on weight loss. Secondary endpoints will evaluate the impact of low fructose diet on blood pressure and cardiovascular biochemical profile.

If fructose is a causal pathway to obesity and metabolic syndrome, it may represent an important target to mitigate this important health problem.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a Body Mass Index (BMI) > 25. BMI defined as: Weight in kilograms divided by Height (squared) in meters.
* Residents of Mexico city
* Healthy individuals (no comorbidities or drug prescription for associated chronic diseases)

Exclusion Criteria:

* Diabetes Mellitus Type 1 or 2
* Severe Hypertension (defined as systolic blood pressure > 160 mmHg and /or diastolic blood pressure > 100 mmHg) and/or Hypertension on pharmacological treatment.
* Chronic Kidney Disease (Glomerular Filtration Rate (GFR) < 60 ml/min)
* Hepatic Damage or Advanced Disease (clinical, biochemical or histological)
* Patient receiving any pharmacological treatments for hypercholesterolemia and/or elevated triglycerides.
* Anemia (any etiology)
* Malignancy
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Somatometry: including weight, height, Body Mass Index (BMI), % Body fat levels, waist and hip index, and blood pressure levels measurements performed by a single evaluator and calibrated equipment | results obtained at the same day of evaluation (weekly monitoring during 6 weeks for each patient)
  measurements will be performed by a trained evaluator

SECONDARY OUTCOMES:
Blood samples: to evaluate metabolic syndrome parameters | basal and final (6 weeks interval between the basal and final results, for each patient)
  samples will be obtained after an eight fasting period

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, MD, Principal Investigator — Instituto Nacional de Cardiología Ignacio Chávez
Locations (1):
- Instituto Nacional de Cardiología Igancio Chávez, Mexico City, Mexico City, Mexico